CLINICAL TRIAL: NCT04805528
Title: Prospective Study of Non-invasive Acupuncture-like Transcutaneous Electrical Nerve Stimulation (Altens) to Help Alleviate Xerostomia After Radiation Therapy for Cancers of the Head and Neck
Brief Title: Study of Non-invasive Acupuncture-like Transcutaneous Electrical Nerve Stimulation (Altens) to Help Alleviate Xerostomia After Radiation Therapy for Cancers of the Head and Neck
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Michael Cummings, Assistant Professor - Department of Radiation Oncology (SMD), University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RHAN20083
Record Dates: First submitted 2021-03-15; First posted 2021-03-18 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Head and Neck Cancer
Keywords: Acupuncture-Like Transcutaneous Electrical Stimulation (ALTENS); Head and Neck Cancer; dry mouth
MeSH Terms: conditions — Head and Neck Neoplasms; Xerostomia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Acupuncture-Like Transcutaneous Electrical Stimulation (ALTENS) Therapy (Experimental): Six (6) small electrodes will be placed on specific points of the body using adhesive pads. These electrodes are connected to the ALTENS device, which will send controlled, low-level electrical impulses through the skin and into the tissue underneath.
  Interventions: Radiation: Acupuncture-Like Transcutaneous Electrical Stimulation (ALTENS)

INTERVENTIONS:
Radiation: Acupuncture-Like Transcutaneous Electrical Stimulation (ALTENS) — Twice weekly ALTENS therapy for 12 weeks

SUMMARY:
The purpose of this study would like to learn if acupuncture-like electrical therapy can be used in patients with head and neck cancer who have had radiation treatment to treat dry mouth.

DETAILED DESCRIPTION:
In this study the investigator would like to better understand if acupuncture-like electrical therapy can be used in patients with head and neck cancer who have had radiation treatment to treat dry mouth. Acupuncture has been shown to help some people with symptoms of dry mouth, and low-level electrical stimulation of acupuncture points has been shown to have similar results as acupuncture treatment with needles.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* No restrictions on gender or ethnicity
* Ability and willingness to present for ALTENS therapy over 12 weeks
* Previous radiation to the head and neck with a dose > 50 Gy
* Subjective complaint of dry mouth
* No evidence of active malignancy in the head and neck region
* Minimum of 3 months post initial curative therapy with no evidence of active disease by standard of care surveillance scans for said disease site

Exclusion Criteria:

* Age under 18 years of age
* Inability to present for ALTENS therapy
* Inability to fill out quality of life questionnaires
* Ability and desire to receive concurrent chemoradiation therapy
* Because ALTENs may stimulate nerves similar to those of pilocarpine, the following exclusions are noted as theoretically ALTENS could produce worse symptoms

  * Unstable Angina
  * Unstable cardiac disease with hospitalization in the last 6 months
  * Presence of a pacemaker, ICD, or other electronic implanted device that could be affected
  * Myocardial infarction in the last 6 months
  * Symptomatic arrhythmia in the last 6 months
  * Severe COPD with exacerbation causing hospitalization within the last 6 months
* Pregnancy or the possibility of pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with a mean parotid dose > 25 Gy have an improvement on the XeQoL questionnaire that is significantly different than those with a mean dose < 25 Gy | 6 Months
  Measure by responses to XeQoL questionnaire

SECONDARY OUTCOMES:
Incidence of Treatment-Related Adverse Events [Safety and Tolerability] | 6 Months
  Measured by adverse event severity and quantity

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No